CLINICAL TRIAL: NCT05535088
Title: Immediate and Short-term Effects in Older Adults With the Use of Virtual Reality
Brief Title: Older Adults Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Ignacio Lassaga, Assistant researcher, University of Gran Rosario
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/20
Record Dates: First submitted 2022-08-26; First posted 2022-09-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Aged

STUDY DESIGN:
Intervention Model Description: The virtual reality will be applied by using a head mounted display. A minute of immersion was repited 6 times
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental): Virtual reality
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Virtual reality consists for about a minute and a half 6 times per session. During the first and the second session, subjects will experiment virtual reality while sited. Moreover, during the third and the fourth session subjects will be standing with a side by side stand. During the last two experimental sessions subjetcts will be standing with a semi tandem stand.

SUMMARY:
In the older adult population, over the years, progressive changes are generated on the different functions and systems of the human body. The musculoskeletal system is not exempt from this process, with the loss of muscle associated with aging being one of the main problems for the older adult population. These alterations bring with them a decrease in muscle strength, along with a loss of functional capacity. Among all the consequences that these deficits can generate, there are: alterations in gait, difficulties in daily transfers, alterations in balance, among others. These changes develop as a consequence an increased risk of falling, these being one of the main causes of morbidity and mortality in the elderly.

As technological development advances, new devices are being created that allow new forms of training our senses and abilities. Since its conception, in the late 1980s, virtual reality has been an area of growing possibilities. Butler and Willet define virtual reality as a technology that allows the user to interact directly with a computer-simulated environment. This tool is gaining more and more interest in the motor rehabilitation of multiple pathologies and also as an option for stability training in older patients. The aim of this study is to evaluate changes in stability after a 2 weeks protocol of virtual reality

DETAILED DESCRIPTION:
This is a quasi-experimental study with a sample of 35 volunteers. Patients of both genders and over 60 years old will be potential candidates for participating in the study. Volunteers will be invited to participate in the study through social networks and e-mail.

The study will be conducted in 6 experimental sessions on different days and 2 assessment days. During assessment sessions several measurements will be performed, including: balance (will be assessed using a balance tracking system balance plate) function (will be assessed by using the Short Physical Performance Battery) and cybersikness (will be assessed using the Sickness Simulator Questionnaire).

The experimental sessions consist in virtual reality immersion for about 1 minute 6 times per session. During the first and the second session, subjects will experiment virtual reality while sited. Moreover, during the third and the fourth session subjects will be standing with a side by side stand. During the last two experimental sessions subjects will be standing with a semi tandem stand.

The one-tailed a priori sample size calculation used the effect size calculated to detect 2.39 cm2 of difference in the displacement area parameter. The sample size for the study was calculated as α set at 5% and the expected power (1-β) at 95%. The analysis returned a minimal sample of 35 participants. With an actual power of 0.95. The G-Power (v. 3.1.9.7, Franz Faul, University Kiel, Germany).

ELIGIBILITY:
Inclusion Criteria:

To have signed the informed consent.

Exclusion Criteria:

* Surgical history of the lower extremities
* Uncontrolled neurological, metabolic, cardiac or respiratory disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Change in balance | At baseline and 2 weeks later
  Balance will be assessed using a balance tracking system balance plate (Balance Tracking Systems, San Diego, CA). Participants stood on the plate for six testing trials. The first three measurement were made with bipedal stance and eyes closed, for about 30 seconds. The next three assessments were made with monopodal support on the right foot and the las 3 measurements were made with monopodal support on the left foot each monopodal repetition last 15 seconds.

SECONDARY OUTCOMES:
Function | At baseline and 2 weeks later
  The function was assessed by using the Short Physical Performance Battery. This is a series of 3 tests to assess lower extremity physical function: a 4-meter walk at usual pace, time to complete 5 unassisted chair stands, and 3 standing balance tests. The scores range from 0 (worst performance) to 12 (best performance).
Change in cybersikness | First day and 2 weeks later
  Cybersickness was assessed by using the "Sickness Simulator Questionnaire" wich consists in 16 questions.
Handgrip | Baseline
  The handgrip was assessed using a Jamar dynamometer while the subjects were sited.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina